CLINICAL TRIAL: NCT00451373
Title: Acute Renal Failure in the Surgical Intense Care Units - NTUH-SICU-ARF (NSARF) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 9561709099; 31MD03
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2007-01

CONDITIONS: Acute Renal Failure; Sepsis; Postoperative
Keywords: ARF, dialysis, cytokine, free radical, major operations
MeSH Terms: conditions — Acute Kidney Injury; Sepsis | interventions — Vancomycin; Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CVVH and SLED
Drug: Vancomycin
Drug: Daptomycin
Device: FX60, AV600 (dialyzer)

SUMMARY:
We examine the prognosis and etiology of postoperative acute renal failure

DETAILED DESCRIPTION:
Postoperative acute renal failure is a serious complication resulting in a prolonged stay and high mortality. Acute renal failure (ARF) develops in 5 to 30% of patients who undergo surgery, and for all causes, it is associated with mortality rates of 60-90%. Despite advances in supportive care and innovations in renal replacement therapies over the past three decades, the mortality rate for these patients remains high. In the previous analysis of NSARF (National Taiwan University Hospital-Surgical Intense Care Unit- acute renal failure database), the mortality rate of acute renal failure patients in SICU is 66.4%, dialysis dependent rate after ARF is 5% and renal recovery rate is 28.6%. Therefore, the issue concerned is to increase the survival rate and renal recovery rate after acute renal failure.

Perioperative ischemic reperfusion injury may result in acute renal failure (ARF), from which patients can invariably recover. However, there remains a large number of patients whose kidneys fail to recover from ARF, and therefore long-term dialysis is required. The dys-regulation of the inflammatory response in critically ill patients has been implicated as an important mechanism underlying the development of multiple organ system dysfunction, septic shock, and death. Furthermore, an increase in oxidative stress is considered an important pathogenic mechanism in the development of ischemic and toxic renal tubular injury. We hypothesize that extensive immune dys-regulation and increased oxidative stress might be an important factor leading to ARF, and/or associated with their all-cause mortality in critically ill patients.

In this study, we will find out (1) first year, the relationship between cytokine storm and free radical storm with urine output during post-surgical ARF, and the effect of renal replacement therapy on serum cytokines and free radical level (2) 2nd year, the difference outcome between low low-efficient daily dialysis (SLEDD), and low low-efficient daily dialysis-hemofiltration (SLEDD-f), the pharmacokinetics of the SLEDD (3) the 3rd year, we sill established the disease severity score of post-operative ARF patients. (NSARF score) and focus on long-term outcomes for survivors of postoperative ARF. From diagnosis to prognosis, we will incorporate important markers of disease diagnosis, treatment and long term outcome. Finally, we hope to improve the mortality and the life quality of postoperative ARF.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative acute renal failure

Exclusion Criteria:

* Patients with ECMO or IABP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2006-07; Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
the mortality of postoperative acute renal failure

SECONDARY OUTCOMES:
the cytokine and free radical change of postoperative renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, MD, PhD, Principal Investigator — National Taiwan University Hosptial; VinCent Wu, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Marshall MR, Golper TA, Shaver MJ, Alam MG, Chatoth DK. Sustained low-efficiency dialysis for critically ill patients requiring renal replacement therapy. Kidney Int. 2001 Aug;60(2):777-85. doi: 10.1046/j.1523-1755.2001.060002777.x. PMID 11473662
- [Background] de Mendonca A, Vincent JL, Suter PM, Moreno R, Dearden NM, Antonelli M, Takala J, Sprung C, Cantraine F. Acute renal failure in the ICU: risk factors and outcome evaluated by the SOFA score. Intensive Care Med. 2000 Jul;26(7):915-21. doi: 10.1007/s001340051281. PMID 10990106